CLINICAL TRIAL: NCT06328023
Title: Association of History of Concussion With Sleep and Physical Performance in Contact Sports Athletes
Brief Title: Impact of Concussion History on Sleep and Physical Performance in Contact Sports Athletes
Status: Recruiting | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/MS-PT/01831
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Concussion, Mild; Sleep; Physical Performance
Keywords: Contact sports
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SCOAT 6 to find association — we will use SCOAT 6 to find the association between concussion , sleep and physical performance

SUMMARY:
This study investigates the correlation between a history of concussions and its effects on both sleep patterns and physical performance among athletes engaged in contact sports. By examining the relationship between concussion history, sleep quality, and athletic performance, this research aims to provide insights into the potential long-term implications of concussions on the well-being and performance of athletes in contact sports

DETAILED DESCRIPTION:
This study delves into the intricate relationship between the history of concussions, sleep quality, and physical performance among athletes participating in contact sports. Concussions, often occurring due to the high-impact nature of these sports, have raised concerns regarding their potential long-term effects on athletes' health and performance. This research aims to elucidate whether a history of concussions influences athletes' sleep patterns and subsequently affects their physical performance.

The study employs a comprehensive approach, utilizing both subjective and objective measures to assess sleep quality, such as self-reported sleep disturbances and objective sleep monitoring techniques. Furthermore, various metrics are employed to evaluate physical performance, including agility, strength, speed, and endurance tests tailored to the specific demands of contact sports.

By analyzing the data collected from athletes with and without a history of concussions, the study aims to identify potential correlations between concussion history, sleep disturbances, and diminished physical performance. Additionally, the research seeks to uncover any potential mediating factors, such as psychological distress or neurocognitive deficits, which may contribute to these associations.

The findings of this study hold significant implications for athlete well-being and sports medicine practices. Understanding the impact of concussions on sleep quality and physical performance can inform tailored interventions and rehabilitation strategies to mitigate the adverse effects of concussions on athletes' health and optimize their performance outcomes in contact sports. Moreover, these insights may contribute to the development of preventive measures and policies aimed at reducing the incidence and severity of concussions in sports settings.

ELIGIBILITY:
Inclusion Criteria:

Participants falling in this category would be recruited into the study.

* Active Male Combat sports player.
* Age between 18-25 years.
* Athletes who had a hit on jaw, neck, head and had symptom of concussion discussed under heading of Introduction.
* Athlete who had history of concussion between 3-30 days.
* Mild concussion according to CANTU NO LOC PTA

Exclusion Criteria:

Participants fall in this category would be excluded of the study.

* Concussion other than sports.
* History of metabolic diseases.
* History of recent fractures

Ages: 18 Years to 36 Years | Sex: All
Age Groups: Adult
Study Population: The athletes will be from contact sports s they are more prone to concussion
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
Cantu Scale | 3 -30 DAYS
  First we have to identify mild concussion which can be done by CANTU SCALE DEVELOPED BY DR ROBER CANTU It has following description In Grade 1 concussions, there may be brief confusion or disorientation immediately following the injury, but there is no loss of consciousness or post-traumatic amnesia. Symptoms resolve within 15 minutes.(MODERATE) Grade 2 concussions involve a loss of consciousness lasting less than one minute and post-traumatic amnesia lasting less than 24 hours. Symptoms, however, persist for more than 15 minutes.(MILD) This is the most severe grade on the Cantu Scale. Grade 3 concussions involve a loss of consciousness lasting more than one minute, post-traumatic amnesia lasting more than 24 hours, and symptoms that persist for more than seven days.(SEVERE)

SECONDARY OUTCOMES:
Sport Concussion Office Assessment Tool 6 | 3 to 30 days
  The SCOAT6 (Sport Concussion Assessment Tool 6) can be used for diagnosis, evaluation, management, and referral for sports-related concussions. It includes:
  History Global symptom scale total symptom number 25 symptom severity 25x6 Verbal Cognitive Test Months in Reverse Order Vital Signs Monitoring Cervical Spine Assessment Neurological Examination Balance Assessment: BESS total 30 10 forrorr each task and score 1 for 1 error Modified Vestibular/Ocular-Motor Screening (mVOMS): 0 -10 4 maybe concussed Anxiety(GAD-7), Depression(PHQ-2), and Sleep Screening ASSQ
  \Graded Exercise Protocols

CONTACTS AND LOCATIONS:
Overall Officials: Nadia ishtiaq, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- HAYATABAD Sports complex, Peshawar, Khyber Pakhtun Khawan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arliani GG, Astur DC, Yamada RK, Yamada AF, da Rocha Correa Fernandes A, Ejnisman B, de Castro Pochini A, Cohen M. Professional football can be considered a healthy sport? Knee Surg Sports Traumatol Arthrosc. 2016 Dec;24(12):3907-3911. doi: 10.1007/s00167-015-3636-2. Epub 2015 May 17. PMID 25982623
- [Background] Hall Z, Baxter G, Dong NX, Chou S-F. Prevention Strategies of Traumatic Brain Injury in Football Players. 2018
- [Background] Sisodia V, Hamid J, Guru K. Efficacy of vestibular rehabilitation in management of balance deficit in Indian collegiate football players, with sport-related concussion-randomized clinical trial. Physiotherapy. 2015;101:e1403-e4.
- [Background] Park E, Baker AJ. Translational Mild Traumatic Brain Injury Research: Bridging the Gap Between Models and Clinical Uncertainty. Neurotrauma: A Comprehensive Textbook on Traumatic Brain Injury and Spinal Cord Injury. 2018:271.
- [Background] Gasquoine PG. Historical perspectives on evolving operational definitions of concussive brain injury: From railway spine to sport-related concussion. Clin Neuropsychol. 2020 Feb;34(2):278-295. doi: 10.1080/13854046.2019.1621383. Epub 2019 May 31. PMID 31146639
- [Background] Broglio SP, Collins MW, Williams RM, Mucha A, Kontos AP. Current and emerging rehabilitation for concussion: a review of the evidence. Clin Sports Med. 2015 Apr;34(2):213-31. doi: 10.1016/j.csm.2014.12.005. Epub 2015 Jan 24. PMID 25818710
- [Background] Clark MD, Asken BM, Marshall SW, Guskiewicz KM. Descriptive Characteristics of Concussions in National Football League Games, 2010-2011 to 2013-2014. Am J Sports Med. 2017 Mar;45(4):929-936. doi: 10.1177/0363546516677793. Epub 2017 Jan 5. PMID 28056179
- [Background] O'Connor KL, Rowson S, Duma SM, Broglio SP. Head-Impact-Measurement Devices: A Systematic Review. J Athl Train. 2017 Mar;52(3):206-227. doi: 10.4085/1062-6050.52.2.05. PMID 28387553
- [Background] Collins MW, Sandel N, Norwig JA, Ruef S. Sport-related Concussion: Experience from the National Football League. Return to Play in Football: Springer; 2018. p. 699-711.
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Alsalaheen BA, Mucha A, Morris LO, Whitney SL, Furman JM, Camiolo-Reddy CE, Collins MW, Lovell MR, Sparto PJ. Vestibular rehabilitation for dizziness and balance disorders after concussion. J Neurol Phys Ther. 2010 Jun;34(2):87-93. doi: 10.1097/NPT.0b013e3181dde568. PMID 20588094
- [Background] McCrea M, Guskiewicz KM, Marshall SW, Barr W, Randolph C, Cantu RC, Onate JA, Yang J, Kelly JP. Acute effects and recovery time following concussion in collegiate football players: the NCAA Concussion Study. JAMA. 2003 Nov 19;290(19):2556-63. doi: 10.1001/jama.290.19.2556. PMID 14625332
- [Background] Balatsouras DG, Koukoutsis G, Aspris A, Fassolis A, Moukos A, Economou NC, Katotomichelakis M. Benign Paroxysmal Positional Vertigo Secondary to Mild Head Trauma. Ann Otol Rhinol Laryngol. 2017 Jan;126(1):54-60. doi: 10.1177/0003489416674961. Epub 2016 Oct 25. PMID 27780909
- [Background] Murray DA, Meldrum D, Lennon O. Can vestibular rehabilitation exercises help patients with concussion? A systematic review of efficacy, prescription and progression patterns. Br J Sports Med. 2017 Mar;51(5):442-451. doi: 10.1136/bjsports-2016-096081. Epub 2016 Sep 21. PMID 27655831
- [Background] Gurr B, Moffat N. Psychological consequences of vertigo and the effectiveness of vestibular rehabilitation for brain injury patients. Brain Inj. 2001 May;15(5):387-400. doi: 10.1080/02699050010005904. PMID 11350653
- [Background] Hoffer ME, Gottshall KR, Moore R, Balough BJ, Wester D. Characterizing and treating dizziness after mild head trauma. Otol Neurotol. 2004 Mar;25(2):135-8. doi: 10.1097/00129492-200403000-00009. PMID 15021772
- [Background] Bell DR, Guskiewicz KM, Clark MA, Padua DA. Systematic review of the balance error scoring system. Sports Health. 2011 May;3(3):287-95. doi: 10.1177/1941738111403122. PMID 23016020